CLINICAL TRIAL: NCT02257918
Title: A Randomized, Open-label Phase 2 Study to Evaluate the Efficacy and Safety of a Single Dose of Oral AZD0914 Compared to Intramuscular Ceftriaxone in the Treatment of Male and Female Subjects With Uncomplicated Gonorrhea
Brief Title: Randomized, Open-label Phase 2 Study of Oral AZD0914 in the Treatment of Gonorrhea
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Purpose: Treatment
Other Study IDs: 14-0014; HHSN272201300012I
Record Dates: First submitted 2014-09-19; First posted 2014-10-07 (Estimated); Results first posted 2017-02-08 (Estimated); Last update posted 2017-03-22 (Actual); Status verified 2016-01-05

CONDITIONS: Gonorrhoea
Keywords: antibiotic; antimicrobial; AZD0914; Ceftriaxone; drug-resistant; sexually transmitted infection; urogenital gonorrhoea
MeSH Terms: conditions — Gonorrhea; Sexually Transmitted Diseases | interventions — zoliflodacin; Ceftriaxone

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group 1 (Experimental): N = 70 subjects receive single oral dose , 2000 mg of AZD0914
  Interventions: Drug: AZD0914
- Group 2 (Experimental): N =70 subjects receive single oral dose , 3000 mg of AZD0914
  Interventions: Drug: AZD0914
- Group 3 (Active Comparator): N = 40 subjects receive single intramuscular dose, 500 mg of ceftriaxone
  Interventions: Drug: Ceftriaxone

INTERVENTIONS:
Drug: AZD0914 — AZD0914 is an antimicrobial amorphous nonsterile powder. Group 1 receive 2000 mg; Group 2 receive 3000 mg. The drug name is also known as ETX0914.
  Arms: Group 1; Group 2
Drug: Ceftriaxone — Ceftriaxone is a broad-spectrum cephalosporin antibiotic with a very long half-life and high penetrability to meninges, eyes and inner ears. A white to yellowish orange crystalline powder. Group 3 receives 500 mg reconstituted with 1 ml Lidocaine HCL 1%, intramuscularly.
  Arms: Group 3

SUMMARY:
This is a multi-center Phase 2 randomized, open-label study in approximately 180 adult male and female subjects, between the ages of 18 and 55, who are in good health and meet all eligibility criteria. The study is designed to assess the safety and efficacy of an antimicrobial investigational product, AZD0914 manufactured by AstraZeneca, administered to adults to treat uncomplicated urogenital gonorrhea compared to treatment with ceftriaxone. Subjects will be randomly assigned 70:70:40 to receive a single, oral dose of 2000 mg of AZD0914, 3000 mg of AZD0914, or intramuscular dose of 500 mg of ceftriaxone. The drug name is also known as ETX0914.

DETAILED DESCRIPTION:
Uncomplicated gonorrhea is currently the second most common bacterial sexually transmitted infection (STI) worldwide and, accordingly, is a serious public health problem. This is a multi-center Phase 2 randomized, open-label study in approximately 180 adult male and female subjects, between the ages of 18 and 55, with uncomplicated cervical or urethral gonorrhea. The study is designed to assess the safety and efficacy of an antimicrobial investigational product, AZD0914 manufactured by AstraZeneca, administered to adults to treat uncomplicated urogenital gonorrhea compared to treatment with intramuscular ceftriaxone. Subjects will be randomly assigned 70:70:40 to receive a single, oral dose of 2000 mg of AZD0914, 3000 mg of AZD0914, or intramuscular dose of 500 mg of ceftriaxone. The study duration is 11 months and subject participation of 30 days. Subjects with 1) untreated urethral or cervical gonorrhea identified via laboratory testing at a prior visit, or 2) untreated subjects acknowledging anal, oral, or vaginal sexual contact in the past 14 days with someone diagnosed with gonorrhea, or 3) signs and symptoms of urethral or cervical gonorrhea will be offered enrollment in the study and consented. The primary objective assess the efficacy by microbiological cure rate of 2000 mg or 3000 mg AZD0914 compared to 500 mg ceftriaxone for the treatment of uncomplicated urogenital gonorrhea. The second primary objective assess the safety and tolerability of a single oral dose of 200 mg or 3000 mg AZD0914 compared to 500 mg ceftriaxone in adult subjects with uncomplicated urogenital gonorrhea. The drug name is also known as ETX0914.

ELIGIBILITY:
Inclusion Criteria:

1. Untreated subjects with signs and symptoms of urethral or cervical gonorrhea, or confirmed urethral or cervical gonorrhea* or any type of sexual contact in the past 14 days with an infected individual. *As defined by positive culture, NAAT test, or Gram-stain 2. Subject is able to give voluntary written informed consent before any study related procedure is performed 3. Willingness to comply with all protocol requirements 4. Male or non-pregnant female 18 to 55 years of age, inclusive 5. If the subject is female, a negative urine pregnancy test at Visit 1 prior to receiving study drug 6. Subject willing to abstain from anal, oral, and vaginal sexual intercourse or use condoms for 7 days following study drug dosing to prevent potential gonococcal reinfection 7. Male subjects must be surgically sterilized or use condoms for 7 days following study drug dosing 8. Female subject must be of non-childbearing potential* or if of childbearing potential, she must be using a highly effective method of birth control** *Non-childbearing potential is defined as being post-menopausal for at least two years, status after bilateral oophorectomy or status after hysterectomy. **Female subjects must avoid becoming pregnant by using one of the following acceptable methods of birth control for 30 days prior to study drug dosing: --Intrauterine contraceptive device; OR --Oral contraceptives; OR --Implanon®,Nexplanon®, DepoProvera®, contraceptive skin patch or NuvaRing®, OR --Tubal ligation OR --Abstinence AND --for 30 days following dosing, any method above should be used plus the required use of a barrier method (condom) by the male partner (even if vasectomized)

Exclusion Criteria:

1. Confirmed or suspected, complicated or systemic gonorrhea such as pelvic inflammatory disease, testicular pain, epididymitis, arthritis, conjunctivitis or endocarditis or clinical proctitis. 2. Known concomitant infection which would require immediate additional systemic antibiotics 3. Female subject currently breastfeeding 4. Use of any systemic or intravaginal antibiotics with activity against N. gonorrhoeae or systemic antivirals within 30 days prior to study drug administration (topical and intravaginal antifugals are permitted). 5. Use of systemic corticosteroid drugs or other immunosuppressive therapy within 30 days prior to enrollment 6. Cytotoxic chemotherapy or radiation therapy within the previous 3 months 7. Known chronic renal, hepatic (including chronic hepatitis B or hepatitis C infection) or hematologic impairment, or other condition that could interfere with the absorption or metabolism of study drug 8. Any concomitant condition that, in the opinion of the Investigator, would preclude an evaluation of a response or make it unlikely that the course of therapy and follow-up could be completed 9. Subject HIV-infected and taking antiretroviral medication -- Subject not HIV-infected and taking antiretroviral for pre- or post- exposure prophylaxis -- Subject newly diagnosed with HIV infection or known to be HIV infected with evidence of immunosuppression, such as documented or patient reported CD4 count of < 200 10. Known allergy to cephalosporin or penicillin antibiotics 11. Receipt or planned receipt of an investigational product in a clinical trial within 30 days prior to or 7 days after study dose administration 12. Female subject is not willing to defer treatment for bacterial vaginosis until Visit 2 if she tests positive for bacterial vaginosis at Visit 1. 13. Use of drugs that act as inducer/inhibitors of CYP3A4/5 or the P-gp efflux transporter* within 30 days prior to study drug administration *such as itraconozale, fluconazole, ketoconazole, verapamil, diltiazem, amiodarone, felodipine, carbamazepine, phenytoin, or St. John's wort 14. Subjects known to be co-infected with chlamydia prior to study entry 15. Subjects with medically documented cardiac arrhythmia 16. Known allergy to lidocaine (or local anesthetics of the amide type, e.g., articaine, bupivacaine, mepivacaine, prilocaine, ropivacaine) or the antimicrobial preservative methylparaben.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 180 (Actual)
Dates: Start 2014-11-25; Primary Completion 2015-12-30 (Actual); Study Completion 2015-12-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Jefferson County Department of Health - STD Clinic, Birmingham, Alabama
  - Indiana University - Bell Flower Clinic, Indianapolis, Indiana
  - CrescentCare Health and Wellness Center, New Orleans, Louisiana
  - Durham County Health Department, Durham, North Carolina
  - Public Health STD Clinic, Seattle, Washington

REFERENCES:
- [Derived] Taylor SN, Marrazzo J, Batteiger BE, Hook EW 3rd, Sena AC, Long J, Wierzbicki MR, Kwak H, Johnson SM, Lawrence K, Mueller J. Single-Dose Zoliflodacin (ETX0914) for Treatment of Urogenital Gonorrhea. N Engl J Med. 2018 Nov 8;379(19):1835-1845. doi: 10.1056/NEJMoa1706988. PMID 30403954

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Untreated participants with signs and symptoms of urethral or cervical gonorrhea, or confirmed urethral or cervical gonorrhea as defined by positive culture, NAAT test, or Gram-stain or any type of sexual contact in the past 14 days with an infected individual were enrolled between 25NOV2014 and 02DEC2015.
Groups:
- AZD0914/ETX0914 2000mg: Participants receive single oral dose of 2000 mg of AZD0914/ETX0914.
- AZD0914/ETX0914 3000mg: Participants receive single oral dose of 3000 mg of AZD0914/ETX0914.
- Ceftriaxone 500mg: Participants receive single intramuscular dose of 500 mg of ceftriaxone.
Period: Overall Study
Arm/Group | AZD0914/ETX0914 2000mg | AZD0914/ETX0914 3000mg | Ceftriaxone 500mg
Started | 72 | 67 | 41
Test of Cure Visit | 72 | 67 | 40
Completed | 68 | 66 | 39
Not Completed | 4 | 1 | 2
Not completed — Lost to Follow-up | 4 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1
Not completed — Pregnancy | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: All participants enrolled and randomized are included in the baseline analysis population.
Groups:
- Total: Total of all reporting groups
Arm/Group | AZD0914/ETX0914 2000mg | AZD0914/ETX0914 3000mg | Ceftriaxone 500mg | Total
Number analyzed (Participants) | 72 | 67 | 41 | 180
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 72 | 67 | 41 | 180
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.2 (8.9) | 28.3 (7.6) | 29.1 (8.2) | 28.8 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 8 | 3 | 13
  Male | 70 | 59 | 38 | 167
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 4 | 4 | 13
  Not Hispanic or Latino | 67 | 63 | 37 | 167
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 1
  Asian | 1 | 2 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 1
  Black or African American | 44 | 40 | 23 | 107
  White | 24 | 19 | 15 | 58
  More than one race | 2 | 5 | 2 | 9
  Unknown or Not Reported | 0 | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 72 | 67 | 41 | 180
Positive culture result for N. gonorrhoeae [Count of Participants; unit: Participants] | 57 | 56 | 28 | 141

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Microbiological Cure at Urethral or Cervical Sites in Each Study Arm
Description: Microbiological cure was assessed at the Test of Cure visit (TOC). Microbiological Cure was derived from the Neisseria gonorrhoeae culture result and assessed by anatomical site. Male participants were swabbed at the urethral site and female participants at the cervical site. Remel RapID NH tests were performed on pure cultures obtained from swab specimens. A participant was defined as a microbiological cure if N. gonorrhoeae was not detectable by culture at TOC.
Time Frame: Day 6
Population: The analysis population was restricted to participants who had a positive culture result for N. gonorrhoeae at the urethral/cervical site at baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | AZD0914/ETX0914 2000mg | AZD0914/ETX0914 3000mg | Ceftriaxone 500mg
Number analyzed (Participants) | 57 | 56 | 28
Participants | 55 | 54 | 28

2. Primary Outcome: Number of Participants Reporting Adverse Events (AEs) and Serious Adverse Events (SAEs) Considered Product-related.
Description: Adverse events are defined as any untoward medical occurrence regardless of its causal relationship to the study treatment. Serious adverse events included any untoward medical occurrence that resulted in death; was life threatening; was a persistent/significant disability/incapacity; required inpatient hospitalization or prolongation thereof was a congenital anomaly/birth defect; or may have jeopardized the subject or required intervention to prevent one of the outcomes. Relationship to study product was determined by the investigator and defined as a reasonable possibility that the study product caused the adverse event. Reasonable possibility means that there is evidence to suggest a causal relationship between the study product and the adverse event.
Time Frame: Day 1 through Day 31
Population: All participants who received the study treatment were included in the analysis population. One participant enrolled in the Ceftriaxone arm was pregnant at enrollment and therefore, not treated.
Measure: Count of Participants; unit: Participants
Arm/Group | AZD0914/ETX0914 2000mg | AZD0914/ETX0914 3000mg | Ceftriaxone 500mg
Number analyzed (Participants) | 72 | 67 | 40
Participants
  Related AEs | 9 | 12 | 6
  Related SAEs | 0 | 0 | 0

3. Secondary Outcome: Number of Participants With Microbiological Cure at Rectal Sites in Each Study Arm
Description: Microbiological cure was assessed at the TOC visit. Microbiological cure was derived from the Neisseria gonorrhoeae culture result and assessed by anatomical site. All participants were swabbed at the rectal site. Remel RapID NH tests were performed on pure cultures obtained from swab specimens. A subject was defined as a microbiological cure if N. gonorrhoeae was not detectable by culture at TOC.
Time Frame: Day 6
Population: The analysis population was limited to participants who had a positive culture result at the rectal site for N. gonorrhoeae at baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | AZD0914/ETX0914 2000mg | AZD0914/ETX0914 3000mg | Ceftriaxone 500mg
Number analyzed (Participants) | 5 | 7 | 3
Participants | 5 | 7 | 3

4. Secondary Outcome: Number of Participants With Microbiological Cure at Pharyngeal Sites in Each Study Arm
Description: Microbiological cure was assessed at the Test of Cure visit (TOC). Microbiological Cure was derived from the Neisseria gonorrhoeae culture result and assessed by anatomical site. All subjects were swabbed at the pharyngeal site. Remel RapID NH tests were performed on pure cultures obtained from swab specimens. A participant was defined as a microbiological cure if N. gonorrhoeae was not detectable by culture at TOC.
Time Frame: Day 6
Population: The analysis population was restricted to participants who had a positive culture result for N. gonorrhoeae at the pharyngeal site at baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | AZD0914/ETX0914 2000mg | AZD0914/ETX0914 3000mg | Ceftriaxone 500mg
Number analyzed (Participants) | 8 | 11 | 4
Participants | 4 | 9 | 4

5. Secondary Outcome: Number of Participants With Clinical Cure in Each Study Arm
Description: A clinical cure was defined as the resolution of all signs and symptoms of gonorrhea (e.g. cervical/vaginal/urethral discharge, dysuria, dyspareunia, vulvovaginal irritation, sore throat) that were present at enrollment with the exception of vaginal discharge due to yeast vaginitis or bacterial vaginosis. A clinical failure was defined by the presence of any sign or symptom of gonorrhea that was also present at enrollment with the exception of vaginal discharge due to yeast vaginitis or bacterial vaginosis. The investigator also submitted his/her determination of whether the participant met or did not meet the criteria for clinical cure (or whether it is unknown if the participant met the criteria). In the event the investigator's assessment of clinical cure did not coincide with the definitions of clinical cure/failure, the investigator's assessment was the final adjudicator.
Time Frame: Day 6
Population: The analysis population was restricted to participants who had a positive culture result for N. gonorrhoeae at any anatomical site and reported signs or symptoms of gonorrhea at baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | AZD0914/ETX0914 2000mg | AZD0914/ETX0914 3000mg | Ceftriaxone 500mg
Number analyzed (Participants) | 57 | 49 | 27
Participants | 52 | 46 | 26

6. Secondary Outcome: Number of Participants With no Detectable N. Gonorrhoeae Nucleic Acid in Urethral/Cervical Specimens in Each Study Arm at Baseline.
Description: Gonorrhea and Chlamydia nucleic acid amplification tests (GC/CT NAAT) were performed at baseline with specimens collected at the cervical/urethral site. Detectable nucleic acid was derived from GC/CT NAAT testing. If N. gonorrhoeae nucleic acid was detected, the result of the test was classified as positive. If no nucleic acid was detected, the result of the test was classified as negative. If a clear result could not be determined for any reason, the result of the test was classified as indeterminate.
Time Frame: Day 1 (Baseline)
Population: The analysis population was restricted to participants who had a positive cervical/urethral culture result for N. gonorrhoeae at baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | AZD0914/ETX0914 2000mg | AZD0914/ETX0914 3000mg | Ceftriaxone 500mg
Number analyzed (Participants) | 57 | 56 | 28
Participants | 0 | 0 | 1

7. Secondary Outcome: Number of Participants With no Detectable N. Gonorrhoeae Nucleic Acid in Urethral/Cervical Specimens in Each Study Arm at Day 6.
Description: Gonorrhea and Chlamydia nucleic acid amplification tests (GC/CT NAAT) were performed at Day 6 with specimens collected at the cervical/urethral site. Detectable nucleic acid was derived from GC/CT NAAT testing. If N. gonorrhoeae nucleic acid was detected, the result of the test was classified as positive. If no nucleic acid was detected, the result of the test was classified as negative. If a clear result could not be determined for any reason, the result of the test was classified as indeterminate.
Time Frame: Day 6
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | AZD0914/ETX0914 2000mg | AZD0914/ETX0914 3000mg | Ceftriaxone 500mg
Number analyzed (Participants) | 57 | 52 | 28
Participants | 48 | 42 | 25

8. Secondary Outcome: Number of Participants With no Detectable N. Gonorrhoeae Nucleic Acid in Rectal Specimens in Each Study Arm
Description: Gonorrhea and Chlamydia nucleic acid amplification tests (GC/CT NAAT) were performed at baseline and Day 6 with specimens collected at the rectal site. Detectable nucleic acid was derived from GC/CT NAAT testing. If N. gonorrhoeae nucleic acid was detected, the result of the test was classified as positive. If no nucleic acid was detected, the result of the test was classified as negative. If a clear result could not be determined for any reason, the result of the test was classified as indeterminate.
Time Frame: Baseline and Day 6
Population: The analysis population was restricted to participants who had a positive rectal culture result for N. gonorrhoeae at baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | AZD0914/ETX0914 2000mg | AZD0914/ETX0914 3000mg | Ceftriaxone 500mg
Number analyzed (Participants) | 5 | 7 | 3
Participants
  Baseline | 0 | 0 | 0
  Day 6 | 5 | 7 | 3

9. Secondary Outcome: Number of Participants With no Detectable N. Gonorrhoeae Nucleic Acid in Pharyngeal Specimens in Each Study Arm
Description: Gonorrhea and Chlamydia nucleic acid amplification tests (GC/CT NAAT) were performed at baseline and Day 6 with specimens collected at the pharyngeal site. Detectable nucleic acid was derived from GC/CT NAAT testing. If N. gonorrhoeae nucleic acid was detected, the result of the test was classified as positive. If no nucleic acid was detected, the result of the test was classified as negative. If a clear result could not be determined for any reason, the result of the test was classified as indeterminate.
Time Frame: Baseline and Day 6
Population: The analysis population was restricted to participants who had a positive pharyngeal culture result for N. gonorrhoeae at baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | AZD0914/ETX0914 2000mg | AZD0914/ETX0914 3000mg | Ceftriaxone 500mg
Number analyzed (Participants) | 8 | 11 | 4
Participants
  Baseline | 0 | 0 | 0
  Day 6 | 2 | 6 | 2

10. Secondary Outcome: Median in Vitro Minimum Inhibitory Concentrations (MIC) Against AZD0914/ETX0914 and Ceftriaxone of Gonococcal Isolates From Culture of Isolates From the Urethral/Cervical Sites at Baseline
Description: For all positive cultures of specimens collected from the urethra or cervix, isolates were collected and tested for antimicrobial susceptibility profiles and the minimum inhibitory concentration (MIC) was determined. MIC was defined as the lowest concentration of an antimicrobial that inhibited the visible growth of a microorganism after overnight incubation. The MIC breakpoint was a chosen concentration of an antibiotic which defines whether a bacterial isolate is susceptible or resistant to the antibiotic. If the MIC was less than or equal to the susceptibility breakpoint, the bacteria was considered susceptible to the antibiotic. If the MIC was greater than this value, the bacteria was considered intermediate or resistant to the antibiotic.
Time Frame: Day 1 (Baseline)
Population: The analysis population includes all participants who had isolates collected and results reported at the timepoint.
Measure: Median (Full Range); unit: µg/mL
Arm/Group | AZD0914/ETX0914 2000mg | AZD0914/ETX0914 3000mg | Ceftriaxone 500mg
Number analyzed (Participants) | 57 | 56 | 27
µg/mL
  AZD0914/ETX0914 | 0.125 [0.008 to 0.250] | 0.093 [0.008 to 0.250] | 0.060 [0.008 to 0.250]
  Ceftriaxone | 0.008 [0.001 to 0.030] | 0.008 [0.001 to 0.060] | 0.004 [0.001 to 0.030]

11. Secondary Outcome: Median in Vitro MIC Against AZD0914/ETX0914 and Ceftriaxone of Gonococcal Isolates From Culture of Isolates From the Urethral/Cervical Sites at Day 6
Description: For all positive cultures of specimens collected from the urethra or cervix, isolates were collected and tested for antimicrobial susceptibility profiles and the MIC was determined. MIC was defined as the lowest concentration of an antimicrobial that inhibited the visible growth of a microorganism after overnight incubation. The MIC breakpoint was a chosen concentration of an antibiotic which defines whether a bacterial isolate is susceptible or resistant to the antibiotic. If the MIC was less than or equal to the susceptibility breakpoint, the bacteria was considered susceptible to the antibiotic. If the MIC was greater than this value, the bacteria was considered intermediate or resistant to the antibiotic.
Time Frame: Day 6
Population: The analysis population includes all participants who had isolates collected and results reported at the timepoint.
Measure: Median (Full Range); unit: µg/mL
Arm/Group | AZD0914/ETX0914 2000mg | AZD0914/ETX0914 3000mg | Ceftriaxone 500mg
Number analyzed (Participants) | 2 | 1 | 0
µg/mL
  AZD0914/ETX0914 | 0.188 [0.125 to 0.250] | 0.060 [0.060 to 0.060] |
  Ceftriaxone | 0.012 [0.008 to 0.015] | 0.001 [0.001 to 0.001] |

12. Secondary Outcome: Median in Vitro MIC Against AZD0914/ETX0914 and Ceftriaxone of Gonococcal Isolates From Culture of Isolates From the Rectal Site at Baseline
Description: For all positive cultures of specimens collected from the rectum, isolates were collected and tested for antimicrobial susceptibility profiles and the MIC was determined. MIC was defined as the lowest concentration of an antimicrobial that inhibited the visible growth of a microorganism after overnight incubation. The MIC breakpoint was a chosen concentration of an antibiotic which defines whether a bacterial isolate is susceptible or resistant to the antibiotic. If the MIC was less than or equal to the susceptibility breakpoint, the bacteria was considered susceptible to the antibiotic. If the MIC was greater than this value, the bacteria was considered intermediate or resistant to the antibiotic.
Time Frame: Day 1 (Baseline)
Population: The analysis population includes all participants who had isolates collected and results reported at the timepoint.
Measure: Median (Full Range); unit: µg/mL
Arm/Group | AZD0914/ETX0914 2000mg | AZD0914/ETX0914 3000mg | Ceftriaxone 500mg
Number analyzed (Participants) | 5 | 6 | 3
µg/mL
  AZD0914/ETX0914 | 0.060 [0.030 to 0.125] | 0.093 [0.060 to 0.250] | 0.125 [0.008 to 0.250]
  Ceftriaxone | 0.004 [0.001 to 0.015] | 0.008 [0.004 to 0.008] | 0.004 [0.004 to 0.008]

13. Secondary Outcome: Median in Vitro MIC Against AZD0914/ETX0914 and Ceftriaxone of Gonococcal Isolates From Culture of Isolates From the Rectal Site at Day 6
Description: as for outcome 12
Time Frame: Day 6
Population: The analysis population includes all participants who had isolates collected and results reported at the timepoint, of which there were none for this anatomical site and timepoint.
Arm/Group | AZD0914/ETX0914 2000mg | AZD0914/ETX0914 3000mg | Ceftriaxone 500mg
Number analyzed (Participants) | 0 | 0 | 0

14. Secondary Outcome: Median in Vitro MIC Against AZD0914/ETX0914 and Ceftriaxone of Gonococcal Isolates From Culture of Isolates From the Pharyngeal Site at Baseline
Description: For all positive cultures of specimens collected from the pharynx, isolates were collected and tested for antimicrobial susceptibility profiles and the MIC was determined. MIC was defined as the lowest concentration of an antimicrobial that inhibited the visible growth of a microorganism after overnight incubation. The MIC breakpoint was a chosen concentration of an antibiotic which defines whether a bacterial isolate is susceptible or resistant to the antibiotic. If the MIC was less than or equal to the susceptibility breakpoint, the bacteria was considered susceptible to the antibiotic. If the MIC was greater than this value, the bacteria was considered intermediate or resistant to the antibiotic.
Time Frame: Day 1 (Baseline)
Population: The analysis population includes all participants who had isolates collected and results reported at the timepoint.
Measure: Median (Full Range); unit: µg/mL
Arm/Group | AZD0914/ETX0914 2000mg | AZD0914/ETX0914 3000mg | Ceftriaxone 500mg
Number analyzed (Participants) | 8 | 11 | 4
µg/mL
  AZD0914/ETX0914 | 0.060 [0.030 to 0.250] | 0.125 [0.008 to 0.250] | 0.093 [0.060 to 0.250]
  Ceftriaxone | 0.008 [0.001 to 0.030] | 0.008 [0.004 to 0.060] | 0.006 [0.002 to 0.060]

15. Secondary Outcome: Median in Vitro MIC Against AZD0914/ETX0914 and Ceftriaxone of Gonococcal Isolates From Culture of Isolates From the Pharyngeal Site at Day 6
Description: as for outcome 14
Time Frame: Day 6
Population: The analysis population includes all participants who had isolates collected and results reported at the timepoint.
Measure: Median (Full Range); unit: µg/mL
Arm/Group | AZD0914/ETX0914 2000mg | AZD0914/ETX0914 3000mg | Ceftriaxone 500mg
Number analyzed (Participants) | 4 | 2 | 0
µg/mL
  AZD0914/ETX0914 | 0.125 [0.060 to 0.250] | 0.093 [0.060 to 0.125] |
  Ceftriaxone | 0.012 [0.004 to 0.030] | 0.012 [0.008 to 0.015] |

ADVERSE EVENTS:
Time Frame: All serious and non-serious adverse events were collected for 30 days after study product administration
Description: One enrolled participant was not subsequently treated and is not included in the number at risk.
Arm/Group | AZD0914/ETX0914 2000mg | AZD0914/ETX0914 3000mg | Ceftriaxone 500mg
Serious Adverse Events (participants affected / at risk) | 0/72 | 1/67 | 0/40
Other Adverse Events (participants affected / at risk) | 6/72 | 12/67 | 11/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AZD0914/ETX0914 2000mg (N=72) | AZD0914/ETX0914 3000mg (N=67) | Ceftriaxone 500mg (N=40)
Gun shot wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | AZD0914/ETX0914 2000mg (N=72) | AZD0914/ETX0914 3000mg (N=67) | Ceftriaxone 500mg (N=40)
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 2 (2) | 3 (3)
Gonorrhea (Infections and infestations) | 1 (1) | 4 (4) | 3 (3)
Headache (Nervous system disorders) | 0 (0) | 6 (6) | 2 (2)
Injection Site Pain (General disorders) | 0/0 (0) | 0/0 (0) | 2 (2) — Only the ceftriaxone arm received the study product via injection.
Urethritis (Infections and infestations) | 1 (1) | 0 (0) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less